CLINICAL TRIAL: NCT01578395
Title: Randomized, Double-blinded, Placebo-controlled, Single Center, and Prospective Phase II Clinical Trial to Analyze the Effects of Antioxidant Agents on DNA Double-strand Breaks in Patients After Radiation-based Cardiac Examinations
Brief Title: Impact of Antioxidant Agents on the Number of DNA Double-strand Breaks After Radiation-based Cardiac Examinations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KEK-ZH-NR: 2010-0352
Record Dates: First submitted 2012-04-12; First posted 2012-04-16 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Focus of the Study: DNA Damage Due to Medical Diagnostic X-ray
MeSH Terms: interventions — Radiation Exposure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- N-acetylcysteine (Experimental): This arm consists of 30 patients who will receive 1200mg n-acetylcysteine dissolved in 50ml NaCl 0.9% iv before either low-dose (10 patients) or high-dose (10 patients) radiation exposure, or no radiation exposure (10 patients)
  Interventions: Radiation: Low-dose radiation exposure; Radiation: High-dose radiation exposure; Other: No radiation exposure
- Ascorbic acid (Experimental): This arm consists of 30 patients who will receive 3000 mg ascorbic acid dissolved in 50 ml NaCl 0.9% iv before either low-dose (10 patients) or high-dose (10 patients) radiation exposure, or no radiation exposure (10 patients)
  Interventions: Radiation: Low-dose radiation exposure; Radiation: High-dose radiation exposure; Other: No radiation exposure
- Sodium Chloride (NaCl) (Placebo Comparator): This arm consists of 30 patients who will receive 50 ml NaCl 0.9% iv before either low-dose (10 patients) or high-dose (10 patients) radiation exposure, or no radiation exposure (10 patients)
  Interventions: Radiation: Low-dose radiation exposure; Radiation: High-dose radiation exposure; Other: No radiation exposure

INTERVENTIONS:
Radiation: Low-dose radiation exposure — what: Cardiac CT; dosage: approx. 2-3 mSv; frequency: once
Radiation: High-dose radiation exposure — what: cardiac catheterization procedures; dosage: approx. 75 mSv; frequency: once
Other: No radiation exposure — Subjects not undergoing any radiation exposure

SUMMARY:
Trial with medicinal products

Recent studies revealed that radiation-based procedures in patients may lead to DNA double-strand breaks in human blood lymphocytes. Additionally, ex vivo studies with human blood lymphocytes have shown a protective effect of antioxidant agents which have been described to decrease the number of DNA double-strand breaks.

This study represents a prospective, double-blinded, randomized, single center, and placebo-controlled phase II clinical trial which analyzes the capability of antioxidant agents to decrease the number of DNA double-strand breaks in human blood lymphocytes in patients undergoing radiation-based cardiac examinations (30 patients with high-dose radiation exposure, 30 patients with low-dose radiation exposure, and 30 subjects without radiation exposure).

A protective effect of antioxidant drugs in patients undergoing radiation-based examinations could therefore change patient management and would provide an important clinical impact.

ELIGIBILITY:
Inclusion criteria:

* Male or Female
* 18-70 years of age
* European origin
* Non-smoker
* 30 patients with high-dose radiation exposure from a cardiac examination
* 30 patients with low-dose radiation exposure from a cardiac examination
* 30 subjects without radiation exposure
* Given written informed consent
* Ability to participate in the study

Exclusion criteria:

* no known intolerance against one of the applied study drugs or against substances used for formulation of one of the study drugs or against other drugs with similar chemical structures as one of the study drugs
* Leukemia
* Lymphoma
* Radio- or chemotherapy
* Severe renal failure (GFR<30 ml/min)
* Positive pregnancy test or lactation
* Radiation-based examination within the last 3 days
* Known glucose-6-phosphate-dehydrogenase deficiency
* Known nephrolithiasis (calciumoxalate calculus)
* Intake of barbiturates, tetracyclines, corticosteroids within the last 4 weeks

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2012-04; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Change in the number of DNA double-strand breaks under influence of antioxidant agents vs. placebo | Baseline blood draw before radiation exposure and follow-up blood draw approx. 30 minutes after radiation exposure
  Potential change (before and after radiation exposure) in the number of DNA double-strand breaks under the influence of n-acetylcystein or ascorbic acid will be measured by qualitative and quantitative immunofluorescence studies (immunofluorescence microscopy and FACS analysis) and will be compared to study patients administered with placebo (using the same quantifiaction tools).

SECONDARY OUTCOMES:
Change in the number of DNA double-strand breaks between n-acetylcysteine and ascorbic acid | Baseline blood draw before radiation exposure and follow-up blood draw approx. 30 minutes after radiation exposure
  Potential change (before and after radiation exposure) in the number of DNA double-strand breaks from patients administered with n-acetylcysteine compared to the number of DNA double-strand breaks from patients administered with ascorbic acid. The change in the number of DNA double-strand breaks will be measured by qualitative and quantitative immunofluorescence studies (immunofluorescence microscopy and FACS analysis).
Change in the number of DNA double-strand breaks between no, low, and high radiation exposure | Baseline blood draw before radiation exposure and follow-up blood draw approx. 30 minutes after radiation exposure
  Potential change (before and after radiation exposure) in the number of DNA double-strand breaks between the different study interventions (low-dose radiation exposure, high-dose radiation exposure, and no radiation exposure). The change in the number of DNA double-strand breaks will be measured by qualitative and quantitative immunofluorescence studies (immunofluorescence microscopy and FACS analysis).

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Kaufmann, MD, Principal Investigator — University Hospital Zurich, Division of Nuclear Medicine
Locations (1):
- University Hospital Zurich, Division of Nuclear Medicine, Zurich, Canton of Zurich, Switzerland